CLINICAL TRIAL: NCT01309269
Title: Non-interventional Study to Investigate the Long Term Effects of MIRCERA in Clinical Routine
Brief Title: Observational Study to Investigate the Long-term Effects of MIRCERA in Clinical Routine
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22911
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will assess the effect of long-term treatment with Mircera (methoxy polyethylene glycol-epoetin beta) in chronic kidney disease patients with renal anemia. Data will be collected from each patient for at least 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with chronic kidney disease (CKD), stages IV and V
* Treatment with Mircera according to label

Exclusion Criteria:

* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease patients treated with Mircera for renal anemia
Sampling Method: Probability Sample
Enrollment: 1083 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lüdenscheid, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this non-interventional study, physician was completely free in his/her decision which participants he/she treated with the medication selected in this study, what dosage was chosen, which diagnostic measures were taken, how the course of treatment was monitored and what accompanying or supplemental medications were prescribed.
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta: Participants received methoxy polyethylene glycol-epoetin beta intravenously or subcutaneously as prescribed by the physician and were observed for 24 months. The actual dose was chosen by the physician and was adjusted as necessary.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Started | 1085
Treated | 978
Completed | 245
Not Completed | 840
Not completed — Adverse Event | 56
Not completed — Withdrawal by Subject | 25
Not completed — Lack of Acceptance | 15
Not completed — Other Erythropoiesis-stimulating Agents | 119
Not completed — Kidney Transplant | 25
Not completed — Administrative Problems | 141
Not completed — Other | 256
Not completed — Other | 1
Not completed — Study Completion Data Not Recorded | 95
Not completed — Enrolled but not Treated | 107

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of methoxy polyethylene glycol-epoetin beta during the study course.
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 978
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (13.9)
Gender [Count of Participants; unit: Participants]
  Female | 428
  Male | 550

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Levels at Monthly Intervals
Description: Hemoglobin levels were measured as grams/deciliter (g/dL).
Time Frame: Prior to Day 1, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24
Population: Effectiveness Population I: all participants for whom at least 1 hemoglobin value was documented after the first application of methoxy polyethylene glycol-epoetin beta during the study course. N (number of participants analyzed) = participants evaluable for this measure. n = participants with hemoglobin values during study period considered.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 926
g/dL
  Prior to Day 1 (n=926) | 11.15 (1.21)
  Month 1 (Day 1-45) (n=802) | 11.31 (1.24)
  Month 2 (Day 46-75) (n=715) | 11.33 (1.23)
  Month 3 (Day 76-105) (n=684) | 11.28 (1.32)
  Month 4 (Day 106-135) (n=685) | 11.28 (1.25)
  Month 5 (Day 136-165) (n=602) | 11.25 (1.22)
  Month 6 (Day 166-195) (n=580) | 11.36 (1.27)
  Month 7 (Day 196-225) (n=541) | 11.30 (1.26)
  Month 8 (Day 226-255) (n=516) | 11.31 (1.25)
  Month 9 (Day 256-285) (n=436) | 11.46 (1.28)
  Month 10 (Day 286-315) (n=423) | 11.40 (1.27)
  Month 11 (Day 316-345) (n=402) | 11.44 (1.31)
  Month 12 (Day 346-375) (n=374) | 11.31 (1.27)
  Month 13 (Day 376-405) (n=351) | 11.29 (1.16)
  Month 14 (Day 406-435) (n=344) | 11.26 (1.16)
  Month 15 (Day 436-465) (n=304) | 11.30 (1.20)
  Month 16 (Day 466-495) (n=272) | 11.37 (1.19)
  Month 17 (Day 496-525) (n=265) | 11.34 (1.27)
  Month 18 (Day 526-555) (n=226) | 11.36 (1.13)
  Month 19 (Day 556-585) (n=213) | 11.28 (1.22)
  Month 20 (Day 586-615) (n=187) | 11.16 (1.16)
  Month 21 (Day 616-645) (n=186) | 11.23 (1.16)
  Month 22 (Day 646-675) (n=167) | 11.38 (1.21)
  Month 23 (Day 676-705) (n=143) | 11.34 (1.13)
  Month 24 (Day 706-735) (n=37) | 11.66 (1.23)

2. Primary Outcome: Percentage of Participants Within Pre-defined Range of Hemoglobin Values
Description: Percentage of participants with hemoglobin values within the following pre-defined ranges is presented: 11-12 gram/deciliter (g/dL), 10-12 g/dL, 11-13 g/dL, and 10-13 g/dL.
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24
Population: Effectiveness Population I. N (number of participants analyzed) = participants evaluable for this measure. n = participants with hemoglobin values during study period considered.
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 802
percentage of participants
  11-12 g/dL: Month 1 (Day 1-45) (n=802) | 37.5
  10-12 g/dL: Month 1 (Day 1-45) (n=802) | 61.6
  11-13 g/dL: Month 1 (Day 1-45) (n=802) | 56.0
  10-13 g/dL: Month 1 (Day 1-45) (n=802) | 80.0
  11-12 g/dL: Month 2 (Day 46-75) (n=715) | 39.0
  10-12 g/dL: Month 2 (Day 46-75) (n=715) | 62.2
  11-13 g/dL: Month 2 (Day 46-75) (n=715) | 58.2
  10-13 g/dL: Month 2 (Day 46-75) (n=715) | 81.4
  11-12 g/dL: Month 3 (Day 76-105) (n=684) | 33.5
  10-12 g/dL: Month 3 (Day 76-105) (n=684) | 58.3
  11-13 g/dL: Month 3 (Day 76-105) (n=684) | 53.1
  10-13 g/dL: Month 3 (Day 76-105) (n=684) | 77.9
  11-12 g/dL: Month 4 (Day 106-135) (n=685) | 35.0
  10-12 g/dL: Month 4 (Day 106-135) (n=685) | 62.6
  11-13 g/dL: Month 4 (Day 106-135) (n=685) | 53.4
  10-13 g/dL: Month 4 (Day 106-135) (n=685) | 81.0
  11-12 g/dL: Month 5 (Day 136-165) (n=602) | 36.2
  10-12 g/dL: Month 5 (Day 136-165) (n=602) | 65.3
  11-13 g/dL: Month 5 (Day 136-165) (n=602) | 53.5
  10-13 g/dL: Month 5 (Day 136-165) (n=602) | 82.6
  11-12 g/dL: Month 6 (Day 166-195) (n=580) | 41.9
  10-12 g/dL: Month 6 (Day 166-195) (n=580) | 64.8
  11-13 g/dL: Month 6 (Day 166-195) (n=580) | 57.1
  10-13 g/dL: Month 6 (Day 166-195) (n=580) | 80.0
  11-12 g/dL: Month 7 (Day 196-225) (n=541) | 39.4
  10-12 g/dL: Month 7 (Day 196-225) (n=541) | 62.8
  11-13 g/dL: Month 7 (Day 196-225) (n=541) | 56.6
  10-13 g/dL: Month 7 (Day 196-225) (n=541) | 80.0
  11-12 g/dL: Month 8 (Day 226-255) (n=516) | 37.8
  10-12 g/dL: Month 8 (Day 226-255) (n=516) | 60.9
  11-13 g/dL: Month 8 (Day 226-255) (n=516) | 56.4
  10-13 g/dL: Month 8 (Day 226-255) (n=516) | 79.5
  11-12 g/dL: Month 9 (Day 256-285) (n=436) | 38.1
  10-12 g/dL: Month 9 (Day 256-285) (n=436) | 58.5
  11-13 g/dL: Month 9 (Day 256-285) (n=436) | 58.5
  10-13 g/dL: Month 9 (Day 256-285) (n=436) | 78.9
  11-12 g/dL: Month 10 (Day 286-315) (n=423) | 39.0
  10-12 g/dL: Month 10 (Day 286-315) (n=423) | 60.8
  11-13 g/dL: Month 10 (Day 286-315) (n=423) | 59.1
  10-13 g/dL: Month 10 (Day 286-315) (n=423) | 80.9
  11-12 g/dL: Month 11 (Day 316-345) (n=402) | 38.3
  10-12 g/dL: Month 11 (Day 316-345) (n=402) | 61.9
  11-13 g/dL: Month 11 (Day 316-345) (n=402) | 57.0
  10-13 g/dL: Month 11 (Day 316-345) (n=402) | 80.6
  11-12 g/dL: Month 12 (Day 346-375) (n=374) | 36.6
  10-12 g/dL: Month 12 (Day 346-375) (n=374) | 60.7
  11-13 g/dL: Month 12 (Day 346-375) (n=374) | 54.8
  10-13 g/dL: Month 12 (Day 346-375) (n=374) | 78.9
  11-12 g/dL: Month 13 (Day 376-405) (n=351) | 37.9
  10-12 g/dL: Month 13 (Day 376-405) (n=351) | 63.2
  11-13 g/dL: Month 13 (Day 376-405) (n=351) | 57.5
  10-13 g/dL: Month 13 (Day 376-405) (n=351) | 82.9
  11-12 g/dL: Month 14 (Day 406-435) (n=344) | 35.8
  10-12 g/dL: Month 14 (Day 406-435) (n=344) | 64.0
  11-13 g/dL: Month 14 (Day 406-435) (n=344) | 54.9
  10-13 g/dL: Month 14 (Day 406-435) (n=344) | 83.1
  11-12 g/dL: Month 15 (Day 436-465) (n=304) | 36.2
  10-12 g/dL: Month 15 (Day 436-465) (n=304) | 64.1
  11-13 g/dL: Month 15 (Day 436-465) (n=304) | 54.3
  10-13 g/dL: Month 15 (Day 436-465) (n=304) | 82.2
  11-12 g/dL: Month 16 (Day 466-495) (n=272) | 34.9
  10-12 g/dL: Month 16 (Day 466-495) (n=272) | 64.0
  11-13 g/dL: Month 16 (Day 466-495) (n=272) | 54.8
  10-13 g/dL: Month 16 (Day 466-495) (n=272) | 83.8
  11-12 g/dL: Month 17 (Day 496-525) (n=265) | 35.8
  10-12 g/dL: Month 17 (Day 496-525) (n=265) | 64.2
  11-13 g/dL: Month 17 (Day 496-525) (n=265) | 52.1
  10-13 g/dL: Month 17 (Day 496-525) (n=265) | 80.4
  11-12 g/dL: Month 18 (Day 526-555) (n=226) | 41.6
  10-12 g/dL: Month 18 (Day 526-555) (n=226) | 67.3
  11-13 g/dL: Month 18 (Day 526-555) (n=226) | 57.5
  10-13 g/dL: Month 18 (Day 526-555) (n=226) | 83.2
  11-12 g/dL: Month 19 (Day 556-585) (n=213) | 37.1
  10-12 g/dL: Month 19 (Day 556-585) (n=213) | 62.4
  11-13 g/dL: Month 19 (Day 556-585) (n=213) | 54.5
  10-13 g/dL: Month 19 (Day 556-585) (n=213) | 79.8
  11-12 g/dL: Month 20 (Day 586-615) (n=187) | 36.9
  10-12 g/dL: Month 20 (Day 586-615) (n=187) | 62.0
  11-13 g/dL: Month 20 (Day 586-615) (n=187) | 54.0
  10-13 g/dL: Month 20 (Day 586-615) (n=187) | 79.1
  11-12 g/dL: Month 21 (Day 616-645) (n=186) | 37.1
  10-12 g/dL: Month 21 (Day 616-645) (n=186) | 63.4
  11-13 g/dL: Month 21 (Day 616-645) (n=186) | 55.4
  10-13 g/dL: Month 21 (Day 616-645) (n=186) | 81.7
  11-12 g/dL: Month 22 (Day 646-675) (n=167) | 47.9
  10-12 g/dL: Month 22 (Day 646-675) (n=167) | 68.3
  11-13 g/dL: Month 22 (Day 646-675) (n=167) | 63.5
  10-13 g/dL: Month 22 (Day 646-675) (n=167) | 83.8
  11-12 g/dL: Month 23 (Day 676-705) (n=143) | 30.8
  10-12 g/dL: Month 23 (Day 676-705) (n=143) | 61.5
  11-13 g/dL: Month 23 (Day 676-705) (n=143) | 54.5
  10-13 g/dL: Month 23 (Day 676-705) (n=143) | 85.3
  11-12 g/dL: Month 24 (Day 706-735) (n=37) | 35.1
  10-12 g/dL: Month 24 (Day 706-735) (n=37) | 54.1
  11-13 g/dL: Month 24 (Day 706-735) (n=37) | 51.4
  10-13 g/dL: Month 24 (Day 706-735) (n=37) | 70.3

3. Primary Outcome: Average Methoxy Polyethylene Glycol-epoetin Beta Dose
Description: Average methoxy polyethylene glycol-epoetin beta dose per application by study month. Mean values were taken when more than 1 application was documented for a participant during the time period considered.
Time Frame: Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24
Population: Effectiveness Population I. N (number of participants analyzed) = participants evaluable for this measure. n = participants with methoxy polyethylene glycol-epoetin beta dose values during study period considered.
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 933
microgram (mcg)
  Month 1 (Day 1-45) (n=933) | 103.23 (68.23)
  Month 2 (Day 46-75) (n=797) | 102.27 (70.96)
  Month 3 (Day 76-105) (n=785) | 102.48 (71.23)
  Month 4 (Day 106-135) (n=758) | 102.64 (70.88)
  Month 5 (Day 136-165) (n=700) | 104.55 (74.81)
  Month 6 (Day 166-195) (n=673) | 102.87 (76.01)
  Month 7 (Day 196-225) (n=631) | 101.08 (77.76)
  Month 8 (Day 226-255) (n=562) | 103.13 (77.41)
  Month 9 (Day 256-285) (n=509) | 103.31 (78.43)
  Month 10 (Day 286-315) (n=481) | 104.62 (77.59)
  Month 11 (Day 316-345) (n=452) | 103.37 (75.16)
  Month 12 (Day 346-375) (n=396) | 104.88 (77.43)
  Month 13 (Day 376-405) (n=382) | 103.63 (79.82)
  Month 14 (Day 406-435) (n=375) | 107.37 (81.52)
  Month 15 (Day 436-465) (n=328) | 105.49 (80.50)
  Month 16 (Day 466-495) (n=290) | 113.21 (82.47)
  Month 17 (Day 496-525) (n=281) | 107.10 (82.63)
  Month 18 (Day 526-555) (n=262) | 101.96 (81.36)
  Month 19 (Day 556-585) (n=230) | 107.25 (80.88)
  Month 20 (Day 586-615) (n=196) | 110.81 (87.95)
  Month 21 (Day 616-645) (n=201) | 107.80 (90.14)
  Month 22 (Day 646-675) (n=166) | 109.98 (88.88)
  Month 23 (Day 676-705) (n=144) | 118.49 (102.60)
  Month 24 (Day 706-735) (n=46) | 116.30 (88.00)

ADVERSE EVENTS:
Time Frame: Day 1 up to Month 24
Description: Safety Analysis Set
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Serious Adverse Events (participants affected / at risk) | 172/978
Other Adverse Events (participants affected / at risk) | 120/978
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=978)
Anaemia (Blood and lymphatic system disorders) | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 5
Angina pectoris (Cardiac disorders) | 3
Aortic valve stenosis (Cardiac disorders) | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 6
Atrial flutter (Cardiac disorders) | 2
Atrioventricular block (Cardiac disorders) | 3
Bradyarrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 5
Cardiac disorder (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 8
Cardiac tamponade (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Coronary artery stenosis (Cardiac disorders) | 2
Mitral valve incompetence (Cardiac disorders) | 1
Mitral valve stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 11
Pericardial effusion (Cardiac disorders) | 1
Tricuspid valve incompetence (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypopituitarism (Endocrine disorders) | 1
Pupils unequal (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal symptom (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2
Diverticular perforation (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 2
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 2
Ileus paralytic (Gastrointestinal disorders) | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Chest pain (General disorders) | 3
Death (General disorders) | 21
Device dislocation (General disorders) | 1
Device malfunction (General disorders) | 1
Disease progression (General disorders) | 1
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 6
Mucosal haemorrhage (General disorders) | 1
Multi-organ failure (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Sudden cardiac death (General disorders) | 8
Systemic inflammatory response syndrome (General disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Biliary dilatation (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Abscess (Infections and infestations) | 2
Brain abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 3
Cytomegalovirus enteritis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Enterobacter bacteraemia (Infections and infestations) | 1
Enterobacter infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Gangrene (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Lobar pneumonia (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Perinephric abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 11
Pneumonia chlamydial (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pyelocystitis (Infections and infestations) | 1
Pyonephrosis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 8
Septic shock (Infections and infestations) | 2
Shunt infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Viral myocarditis (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 9
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 5
Pelvic fracture (Injury, poisoning and procedural complications) | 2
Periorbital haematoma (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 2
Shunt occlusion (Injury, poisoning and procedural complications) | 2
Shunt thrombosis (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1
Blood bicarbonate decreased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood lactic acid increased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
C-reactive protein increased (Investigations) | 2
Haemoglobin decreased (Investigations) | 4
Acidosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Alcohol induced persisting dementia (Nervous system disorders) | 1
Brain injury (Nervous system disorders) | 1
Cerebral amyloid angiopathy (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 5
Cerebrovascular accident (Nervous system disorders) | 4
Convulsion (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 2
Grand mal convulsion (Nervous system disorders) | 2
Hepatic encephalopathy (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 2
Azotaemia (Renal and urinary disorders) | 1
Prerenal failure (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 3
Renal haemorrhage (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3
Diabetic foot (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 1
Immobile (Social circumstances) | 1
Treatment noncompliance (Social circumstances) | 1
Amputation (Surgical and medical procedures) | 1
Aortic valve replacement (Surgical and medical procedures) | 1
Arteriovenous shunt operation (Surgical and medical procedures) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1
Coronary artery bypass (Surgical and medical procedures) | 1
Coronary revascularisation (Surgical and medical procedures) | 1
Heart valve operation (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 2
Hysterectomy (Surgical and medical procedures) | 1
Leg amputation (Surgical and medical procedures) | 2
Parathyroidectomy (Surgical and medical procedures) | 2
Thyroidectomy (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Arteriosclerosis moenckeberg-type (Vascular disorders) | 1
Brachiocephalic vein stenosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 4
Peripheral arterial occlusive disease (Vascular disorders) | 6
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Hemiparesis (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=978)
Anaemia (Blood and lymphatic system disorders) | 2
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Hypertensive heart disease (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1
Hypoparathyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Toxic nodular goitre (Endocrine disorders) | 1
Blindness (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Papilla of vater stenosis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Drug ineffective (General disorders) | 1
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 1
Necrosis (General disorders) | 1
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Thrombosis in device (General disorders) | 2
Unevaluable event (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Bacterial disease carrier (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 5
Bronchitis bacterial (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Colostomy infection (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infective myositis (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 1
Shunt infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 6
Wound infection staphylococcal (Infections and infestations) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Femur fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 6
Post procedural haematoma (Injury, poisoning and procedural complications) | 2
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 2
Shunt aneurysm (Injury, poisoning and procedural complications) | 2
Shunt malfunction (Injury, poisoning and procedural complications) | 3
Shunt occlusion (Injury, poisoning and procedural complications) | 5
Shunt stenosis (Injury, poisoning and procedural complications) | 3
Shunt thrombosis (Injury, poisoning and procedural complications) | 1
Blood calcium abnormal (Investigations) | 1
Blood parathyroid hormone increased (Investigations) | 1
C-reactive protein increased (Investigations) | 3
Endoscopy upper gastrointestinal tract (Investigations) | 1
Haemoglobin abnormal (Investigations) | 6
Haemoglobin decreased (Investigations) | 1
Haemoglobin increased (Investigations) | 1
Neurological examination normal (Investigations) | 1
Volume blood decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid arteriosclerosis (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Facial paresis (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2
Haemorrhage subepidermal (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Dependence on enabling machine or device (Social circumstances) | 2
Aneurysm repair (Surgical and medical procedures) | 2
Angioplasty (Surgical and medical procedures) | 2
Arteriovenous fistula operation (Surgical and medical procedures) | 4
Arteriovenous shunt operation (Surgical and medical procedures) | 4
Cataract operation (Surgical and medical procedures) | 1
Central venous catheter removal (Surgical and medical procedures) | 1
Central venous catheterisation (Surgical and medical procedures) | 1
Choledocholithotomy (Surgical and medical procedures) | 1
Coronary angioplasty (Surgical and medical procedures) | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1
Duodenal sphincterotomy (Surgical and medical procedures) | 1
Haemodialysis (Surgical and medical procedures) | 3
Intra-aortic balloon placement (Surgical and medical procedures) | 1
Laser therapy (Surgical and medical procedures) | 1
Leg amputation (Surgical and medical procedures) | 1
Packed red blood cell transfusion (Surgical and medical procedures) | 1
Parathyroidectomy (Surgical and medical procedures) | 1
Radioactive iodine therapy (Surgical and medical procedures) | 1
Rehabilitation therapy (Surgical and medical procedures) | 1
Skin lesion excision (Surgical and medical procedures) | 1
Skin neoplasm excision (Surgical and medical procedures) | 1
Thrombectomy (Surgical and medical procedures) | 2
Thrombolysis (Surgical and medical procedures) | 1
Vasodilation procedure (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 3
Superior vena cava syndrome (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.